CLINICAL TRIAL: NCT05653531
Title: Significance of Hepatic Biomarkers in the Evaluation of Response to Treatment and Prognosis in Lung Cancer Patients Treated With Immune Checkpoint Inhibitors
Brief Title: Clinical Significance of Hepatic Biomarkers in Lung Cancer Patients Treated With Immune Checkpoint Inhibitors
Acronym: HEPATICI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: PI2021_843_0230
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Immune Checkpoint Inhibitor; Lung Cancer; Liver Biomarkers; Transaminases
Keywords: immune checkpoint inhibitor; Lung Cancer; liver biomarkers; transaminases
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample — Liver blood tests (AST, ALT, PAL, GGT, bilirubin, PT) will be performed before each ICI injection during the first three injections and again at 6 months.

SUMMARY:
Lung cancer is the leading cause of cancer death worldwide. The emergence of immune checkpoint inhibitors (ICIs) has revolutionized the treatment of lung cancer over the past 10 years. Nivolumab, ipilimumab, pembrolizumab, atezolizumab, and durvalumab have been successively approved in non-small cell lung cancer, small cell lung cancer, and pleural mesothelioma. Although the efficacy of ICIs is remarkable in some patients, the objective response rate is only about 20%. The development of predictive biomarkers for treatment response is essential. Non-invasive methods and easily accessible biomarkers at low cost are required.ICIs activate the immune system through the inhibition of checkpoints (PD-L1, PD-1). The immune system and the liver are interconnected and constantly interact through a complex regulatory system. Patients with lung cancer frequently suffer from liver damage, due to metastases, treatments or underlying pathologies. The objective of the study is to evaluate the clinical significance of key liver biomarkers (AST, ALT, PAL, GGT, bilirubin, PT) in patients with lung cancer treated with ICI.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Age > 18 years
* Patient with lung cancer of any histological type
* Initiation of ICI therapy
* Signed consent for the study

Exclusion Criteria:

* Patient with previous ICI treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
basal ALT blood concentration in lung cancer patients treated with ICI determined | one year
  To Identify baseline blood ALT concentration as a predictive liver biomarker of treatment response in lung cancer patients treated with ICI.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No